CLINICAL TRIAL: NCT04663815
Title: The Impact of an Animal-assisted Activity on the Stress Level of Hospitalized Children: a Randomized Trial
Brief Title: The Impact of an Animal-assisted Activity on the Stress Level of Hospitalized Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Stress-HC-VS
Record Dates: First submitted 2020-12-02; First posted 2020-12-11 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Hospitalization in Children

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB arm (Other): Animal-assisted activity intervention on 2nd day of hospitalization, control intervention on the 4th day of hospitalization.
  Interventions: Behavioral: Animal-assisted activity; Other: Control intervention
- BA arm (Other): Control intervention on 2nd day of hospitalization, animal-assisted activity intervention on the 4th day of hospitalization.
  Interventions: Behavioral: Animal-assisted activity; Other: Control intervention

INTERVENTIONS:
Behavioral: Animal-assisted activity — The intervention is an animal-assisted activity consisting of a visit to Villa Samson (a place on the campus of the hospital specifically intended for patients to meet pets), where the child will work with a therapy dog for 1 hour. Under supervision, the animal is stroked and combed by the child, they play games together, the child feeds the animal, etc.
Other: Control intervention — The control intervention reenacts a normal stay in the hospital, so the child spends one hour in the hospital room where the child can play, watch tv, etc.

SUMMARY:
The aim of this research is to study the effect of an animal-assisted activity (AAA) on the stress level of hospitalized children.

DETAILED DESCRIPTION:
A hospitalization is a major stressor in a child's life, which can have negative effects on recovery. It is assumed that animal-assisted interventions can have a positive effect on the level of stress, but this has not yet been sufficiently researched. This study aims to measure a possible effect. Children who are hospitalized will receive an animal-assisted activity. A normal afternoon in their hospital room counts as a control activity. The stress level is measured through saliva cortisol, blood pressure, heart rhythm variability and a visual analogue stress scale.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized in the Universitair Ziekenhuis Brussel
* dutch and/or french speaking.

Exclusion Criteria:

* decreased immunity
* multi-resistant germs
* disturbed diabetes
* fever of unknown origin
* fear of animals
* dogs or cats allergy
* cognitive impairment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in heart rate variability (HVR) | 1 hour
  A marker of the activity of the sympathetic nervous system.
Change in systolic and diastolic blood pressure | 1 hour
  A marker of the activity of the sympathetic nervous system.
Change in saliva cortisol | 1 hour
  A marker of the activity of the hypothalamic - pituitary - adrenal axis.
Change in visual analogue stress scale | 1 hour
  A 10-point scale for patient self-reporting of stress. The scale ranges from 0-10 where 0 indicates a better and 10 indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Campforts, MD, PhD, Principal Investigator
Locations (1):
- UZ Brussel, Jette, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellhammer DH, Wust S, Kudielka BM. Salivary cortisol as a biomarker in stress research. Psychoneuroendocrinology. 2009 Feb;34(2):163-171. doi: 10.1016/j.psyneuen.2008.10.026. Epub 2008 Dec 18. PMID 19095358
- [Background] Gamelin FX, Baquet G, Berthoin S, Bosquet L. Validity of the polar S810 to measure R-R intervals in children. Int J Sports Med. 2008 Feb;29(2):134-8. doi: 10.1055/s-2007-964995. Epub 2007 Jul 5. PMID 17614016
- [Background] Lesage FX, Berjot S, Deschamps F. Clinical stress assessment using a visual analogue scale. Occup Med (Lond). 2012 Dec;62(8):600-5. doi: 10.1093/occmed/kqs140. Epub 2012 Sep 10. PMID 22965867
- [Background] Al-Yateem NS, Banni Issa W, Rossiter R. Childhood stress in healthcare settings: awareness and suggested interventions. Issues Compr Pediatr Nurs. 2015 Jun;38(2):136-53. doi: 10.3109/01460862.2015.1035465. Epub 2015 Apr 28. PMID 25919580
- [Background] Ursin H, Eriksen HR. The cognitive activation theory of stress. Psychoneuroendocrinology. 2004 Jun;29(5):567-92. doi: 10.1016/S0306-4530(03)00091-X. PMID 15041082
- [Background] Nassau JH, Tien K, Fritz GK. Review of the literature: integrating psychoneuroimmunology into pediatric chronic illness interventions. J Pediatr Psychol. 2008 Mar;33(2):195-207. doi: 10.1093/jpepsy/jsm076. Epub 2007 Sep 10. PMID 17848391
- [Background] Michels N, Sioen I, Clays E, De Buyzere M, Ahrens W, Huybrechts I, Vanaelst B, De Henauw S. Children's heart rate variability as stress indicator: association with reported stress and cortisol. Biol Psychol. 2013 Oct;94(2):433-40. doi: 10.1016/j.biopsycho.2013.08.005. Epub 2013 Sep 2. PMID 24007813
- [Background] Vessey JA. Children's psychological responses to hospitalization. Annu Rev Nurs Res. 2003;21:173-201. PMID 12858697